CLINICAL TRIAL: NCT05792033
Title: Multicentric Prospective T1 Urinary Bladder Cancer (ROGUE-1) Registry
Brief Title: Multicentric Prospective T1 Urinary Bladder Cancer Registry
Acronym: ROGUE-1
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, David D'Andrea, MD, Medical University of Vienna
Other Study IDs: 2234/2020
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: T1 Urinary Bladder Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prospective registry — Prospective registry of patients with primary diagnosis of T1 urinary bladder cancer

SUMMARY:
Synopsis Rationale Patients with T1 urinary bladder cancer (UBC) are at high risk for recurrence and progression. However, the prognosis is dependent on several concomitant factors. First and foremost, an accurate diagnosis is imperative for an appropriate disease management. Due to conventional transurethral resection technique, resulting in fragmentation and cauterization of the tissue, the pathological review is often difficult and may result in under or over-staging. A central pathology review of EORTC trial data found only a 43% concordance for T1 tumours compared with staging by a local pathologist. Moreover, risk factors such as concomitant carcinoma in situ (CIS), variant histology (VH) and lymphovascular invasion (LVI) have been associated with even poorer prognosis in patients with T1 UBC. However, there is consistent heterogeneity in reporting these features across studies.

There is an unmet need for a clean prospective dataset on T1 UBC to allow an accurate risk stratification in order to aid clinical decision making.

Study endpoints The primary objective of the study is to prospectively collect data on patients with primary diagnosis of T1 NMIBC in order

* to investigate the therapy failure rates in patients with primary diagnosis of T1 bladder cancer
* to investigate the association of clinico-pathologic features such as LVI, VH and CIS, tumor size and number of tumors with pathologic outcomes.
* to analyze the accuracy of the local pathologist assessment on the evaluation of pathology features such as tumor stage and grade, substaging according to the microscopic and extensive invasion, LVI, VH and CIS.
* to investigate the inter-observer variability among different local pathologist comparing these observations with a central pathology revision performed by expert genitourinary pathologist.
* to develop a clinically applicable risk stratification tool which may guide physicians during patient counselling and decision-making regrading adjuvant therapies or early cystectomy

Methods Patients with primary diagnosis of UBC and scheduled for transurethral resection of bladder at international urology departments will be prospectively recruited. Patients with confirmed diagnosis of T1 UBC will be included in the study All selected patients will be asked to sign a written informed consent and any locally required privacy act document authorization prior to TURB. Furthermore, all patients will be required to provide consent for central pathology revision.

Patients will receive adjuvant treatments (i.e. intravesical therapy or early cystectomy) according to guidelines and clinical standards. All data regarding these treatments will be prospectively collected during the study period or patient death.

The clinical data of patients included in the study will be prospectively collected at each center and saved within an electronic case report form (eCRF) using the Castor platform (Castor www.castoredc.com). After combining the data sets from the different centers, reports will be generated for each variable identifying missing or inconsistent data. Incongruities will be solved before freezing the final database. Protected health information (PHI) will be unavailable to investigators at other sites. Follow-up chart abstractions will occur at 6-month intervals until the patient is deceased, lost to follow-up, or the study is terminated.

Pathologic specimens will be scanned and uploaded to the eCRF to allow a central pathologic revision.

Rationale for patient number Recurrence rates for T1 bladder cancer are estimated to be up to 50% [4]. We plan to include 700 patients in the study. This would allow to detect a 50% failure rate with 4% on either side of the 95% Confidence Interval (proportion 0,50 with 95%CI 0.46-0.54).

Future prospects, dissemination and impact A manuscript will be written and submitted for publication on a scientific journal. Any formal presentation or publication of data collected from this trial will be considered as a joint publication by the investigators.

Studies originating from this registry could potentially change the risk stratification and, therefore, the management of patients with T1 UBC.

ELIGIBILITY:
Inclusion criteria

Subjects must meet all the following inclusion criteria to participate in this study:

* Pathologically confirmed diagnosis of primary T1 bladder cancer
* Diagnosis of primary T1 bladder cancer is confirmed at 2nd look TURB
* Imaging examinations shows no lymph node metastasis or distant metastasis
* Patients who agree to surgery, and will be effected to the standard postoperative management and follow-up treatment in accordance to current guidelines
* In case of persistent T1 bladder cancer at 2nd look TURB, patient can be included only if detrusor muscle is present in the pathologic specimen

Exclusion criteria

* Previous bladder cancer
* Upstaging to MIBC at 2nd look TURB
* Contraindications to surgery (i.e. bladder fibrosis)
* Poor performance status making a surgical intervention too risky
* Life expectancy of less than one year
* Patient refused to participate
* Pregnancy
* Concomitant or history of upper urinary tract urothelial cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary diagnosis of T1 urinary bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapy failure | 2021 to 2028
  Proportion of patients failing intravesical BCG Therapy and undergo radical cystectomy and the proportion of patients treated with upfront radical cystectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria